CLINICAL TRIAL: NCT05133999
Title: Iron, Transferrin and Retinopathy of Prematurity (ROP): Towards New Pathophysiological Mechanisms.
Brief Title: Iron and Retinopathy of Prematurity (ROP)
Acronym: Fer-ROP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation VISIO (Unknown); Fondation Université de Paris (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211233; 2021-A02182 (Other: ID-RCB)
Record Dates: First submitted 2021-11-02; First posted 2021-11-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Retinopathy of Prematurity
Keywords: retinopathy; prematurity; ROP; Iron and transferrin; Preterm infants
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Diseases; Premature Birth | interventions — Transferrin; Ferritins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants: infants born at <31 week's post-menstrual age (PMA) or ≤1250g of birth weight
  Interventions: Biological: Plasma determination of iron, transferrin and ferritin; Other: Fundus Examination by wide field digital imaging camera (PanocamTM camera)

INTERVENTIONS:
Biological: Plasma determination of iron, transferrin and ferritin — Iron, transferrin and ferritin levels in plasma
Other: Fundus Examination by wide field digital imaging camera (PanocamTM camera) — ROP screening using wide field digital retinal imaging according to current recommendations.

SUMMARY:
The purpose of this study is to determine whether increased transferrin saturation in plasma (that reflects iron overload and/or low transferrin) is an independent risk factor for ROP development and severity.

Preterm infants born at <31 week's post-menstrual age (PMA) or ≤1250g of birth weight will be included. Iron parameters in plasma will be measured during the first month of life. Retinopathy of prematurity (ROP) will be screened as currently recommended. The relationship between plasma iron parameters and ROP development and/or severity will be established.

DETAILED DESCRIPTION:
The incidence of ROP, the main cause of vision impairment in children, is increasing parallel to the recent changes in practices targeting higher oxygen saturation in preterm babies in many countries following the publication of five trials that showed higher rates of death with lower oxygen saturations. The main risk factor for ROP development is oxygen excess. Oxygen contributes to the formation of reactive oxygen species and to lipid peroxidation which leads to vasoconstriction, vascular cytotoxicity, and arrest of vascular development causing ischemia of retinal neurons, thereby promoting the development of ROP.

90% of extremely low birth weight infants need red blood cell transfusions (RBCT) due to their immature erythropoiesis, frequent blood sampling and small circulating blood volume. RBCT are a major source of iron overload and ferritin plasma levels may remain elevated for several weeks after transfusions. It has been shown that blood transfusion is a risk factor of ROP in preterm infants. However, whether this relationship is mediated by an increased iron load remains controversial.

Only two studies, conducted before the 2000s, identified plasma iron overload as a risk factor for ROP. These studies with a limited number of patients, showed contradictory results, failing to draw a conclusion.

Excess iron worsens oxidative stress. Iron catalyzes the Fenton reaction which leads to the formation of reactive oxygen species. In addition a transferrin deficiency (the main iron chelator) has been suggested in premature infants. The oxidative stress observed in ROP could therefore be the consequence not only of oxygen therapy but also of iron overload.

The main objective of this study is to determine whether increased transferrin saturation in plasma (that reflects iron overload and/or low transferrin) is an independent risk factor for ROP development and severity.

The secondary aims/objectives are :

* Determine whether low transferrin level in plasma is an independent risk factor for ROP development and severity.
* Determine whether iron parameters imbalance in plasma are a risk factor for other comorbidities in Preterm infants i.e.:
* 1) sepsis
* 2) severe bronchopulmonary dysplasia
* 3) necrotizing enterocolitis (stage 2 or 3)
* 4) cystic periventricular leukomalacia
* 5) grade III or IV intraventricular haemorrhage

Study duration will be 29 months, with an inclusion period of 24 months and a last visit for ROP evaluation at 45 week's post-menstrual age (PMA).

A total of 175 patients should be included: 35 with ROP and 140 without ROP.

ELIGIBILITY:
Inclusion Criteria:

* All infants born at <31 week's post-menstrual age (PMA) or ≤1250g of birthweight
* Admitted at two neonatology departments (level III) from birth
* With non-opposition consent of two parents

Exclusion Criteria:

* Congenital malformation
* Life-threatening condition (not expected to survive more than a few days)
* Absence of health care protection.

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born at <31 weeks' PMA or ≤1250 g of birth weight
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
ROP screening | From 31 to 45 weeks' post menstrual age (PMA) [= (term + 4 weeks of life)].
  Presence of ROP development (any stage / any zone in at least one eye) during follow-up.
Levels of transferrin saturation in plasma at 1 week of life | at 1 week of life
  Blood dosage

SECONDARY OUTCOMES:
Levels of iron | at birth, 2, 3, and 4 weeks of life
  Blood dosage, in µmol/l
Levels of transferrin | at birth, 2, 3, and 4 weeks of life
  Blood dosage, in g/l
Levels of ferritin | at birth, 2, 3, and 4 weeks of life
  Blood dosage, in µg/l
ROP's highest stage | during follow-up about 5 months, up to 45 weeks' PMA
  according to International Classification of Retinopathy of Prematury (ICROP3 classification)
Need of treatment for ROP | during follow-up about 5 months, up to 45 weeks' PMA
  Laser, anti-VEGF injections, surgery
Number of each intervention | during follow-up about 5 months, up to 45 weeks' PMA
  Number of each intervention if a treatment was needed
Death or presence of severe co-morbidities in preterm infant | At 36 weeks' PMA
  death or presence of monitoring :
  1) severe bronchopulmonary dysplasia or 2) necrotizing enterocolitis (stage 2 or 3), or 3) cavitary periventricular leucomalacia or 4) intraventricular haemorrhage (grade III or IV).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra DARUICH, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Elsa KERMOVANT, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Pediatrics and neonatal intensive care department - Cochin hospital - Port Royal Maternity, Paris
  - Ophtalmology department _ Necker Enfants Malades Hospital, Paris
  - Pediatrics and noenatal intensive care department - Necker-Enfants Malades Hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Verdier K, Ulla E, Lofgren S, Fernell E. Children with blindness - major causes, developmental outcomes and implications for habilitation and educational support: a two-decade, Swedish population-based study. Acta Ophthalmol. 2018 May;96(3):295-300. doi: 10.1111/aos.13631. Epub 2017 Nov 23. PMID 29168313
- [Background] Manley BJ, Kuschel CA, Elder JE, Doyle LW, Davis PG. Higher Rates of Retinopathy of Prematurity after Increasing Oxygen Saturation Targets for Very Preterm Infants: Experience in a Single Center. J Pediatr. 2016 Jan;168:242-244. doi: 10.1016/j.jpeds.2015.10.005. Epub 2015 Nov 6. PMID 26548746
- [Background] BOOST II United Kingdom Collaborative Group; BOOST II Australia Collaborative Group; BOOST II New Zealand Collaborative Group; Stenson BJ, Tarnow-Mordi WO, Darlow BA, Simes J, Juszczak E, Askie L, Battin M, Bowler U, Broadbent R, Cairns P, Davis PG, Deshpande S, Donoghoe M, Doyle L, Fleck BW, Ghadge A, Hague W, Halliday HL, Hewson M, King A, Kirby A, Marlow N, Meyer M, Morley C, Simmer K, Tin W, Wardle SP, Brocklehurst P. Oxygen saturation and outcomes in preterm infants. N Engl J Med. 2013 May 30;368(22):2094-104. doi: 10.1056/NEJMoa1302298. Epub 2013 May 5. PMID 23642047
- [Background] Sapieha P, Joyal JS, Rivera JC, Kermorvant-Duchemin E, Sennlaub F, Hardy P, Lachapelle P, Chemtob S. Retinopathy of prematurity: understanding ischemic retinal vasculopathies at an extreme of life. J Clin Invest. 2010 Sep;120(9):3022-32. doi: 10.1172/JCI42142. Epub 2010 Sep 1. PMID 20811158
- [Background] Howarth C, Banerjee J, Aladangady N. Red Blood Cell Transfusion in Preterm Infants: Current Evidence and Controversies. Neonatology. 2018;114(1):7-16. doi: 10.1159/000486584. Epub 2018 Mar 16. PMID 29550819
- [Background] Hesse L, Eberl W, Schlaud M, Poets CF. Blood transfusion. Iron load and retinopathy of prematurity. Eur J Pediatr. 1997 Jun;156(6):465-70. doi: 10.1007/s004310050641. PMID 9208245
- [Background] Dani C, Reali MF, Bertini G, Martelli E, Pezzati M, Rubaltelli FF. The role of blood transfusions and iron intake on retinopathy of prematurity. Early Hum Dev. 2001 Apr;62(1):57-63. doi: 10.1016/s0378-3782(01)00115-3. PMID 11245995
- [Background] Inder TE, Clemett RS, Austin NC, Graham P, Darlow BA. High iron status in very low birth weight infants is associated with an increased risk of retinopathy of prematurity. J Pediatr. 1997 Oct;131(4):541-4. doi: 10.1016/s0022-3476(97)70058-1. PMID 9386655
- [Background] Hirano K, Morinobu T, Kim H, Hiroi M, Ban R, Ogawa S, Ogihara H, Tamai H, Ogihara T. Blood transfusion increases radical promoting non-transferrin bound iron in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2001 May;84(3):F188-93. doi: 10.1136/fn.84.3.f188. PMID 11320046
- [Background] Daruich A, Le Rouzic Q, Jonet L, Naud MC, Kowalczuk L, Pournaras JA, Boatright JH, Thomas A, Turck N, Moulin A, Behar-Cohen F, Picard E. Iron is neurotoxic in retinal detachment and transferrin confers neuroprotection. Sci Adv. 2019 Jan 9;5(1):eaau9940. doi: 10.1126/sciadv.aau9940. eCollection 2019 Jan. PMID 30662950
- [Background] Hellstrom A, Engstrom E, Hard AL, Albertsson-Wikland K, Carlsson B, Niklasson A, Lofqvist C, Svensson E, Holm S, Ewald U, Holmstrom G, Smith LE. Postnatal serum insulin-like growth factor I deficiency is associated with retinopathy of prematurity and other complications of premature birth. Pediatrics. 2003 Nov;112(5):1016-20. doi: 10.1542/peds.112.5.1016. PMID 14595040
- [Background] Luo XQ, Zhang CY, Zhang JW, Jiang JB, Yin AH, Guo L, Nie C, Lu XZ, Deng H, Zhang L. Identification of Iron Homeostasis Genes Dysregulation Potentially Involved in Retinopathy of Prematurity Pathogenicity by Microarray Analysis. J Ophthalmol. 2015;2015:584854. doi: 10.1155/2015/584854. Epub 2015 Oct 18. PMID 26557385